CLINICAL TRIAL: NCT07365176
Title: The Protective Role of High-intensity Interval Exercise Compared With Continuous Moderate Exercise on Glycemia Decrease is More Relevant in Postabsorptive vs. Postprandial State in Adults With Type 1 Diabetes
Brief Title: High-intensity Interval Exercise Compared With Continuous Moderate Exercise on Glycemia in Postabsorptive vs. Postprandial State in Adults With Type 1 Diabetes
Acronym: Interdiab 1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universite du Littoral Cote d'Opale (Other)
Responsible Party: Principal Investigator, Herve DEVANNE, PhD, PhD, Universite du Littoral Cote d'Opale
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: IRB00012476-2023-08-02-225
Record Dates: First submitted 2025-12-28; First posted 2026-01-26 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Diabetes Mellitus, Type 1
Keywords: Blood glucose; Exercise; Hypoglycemia
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Motor Activity; Hypoglycemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- A/B/C/D (Experimental): A= High-intensity interval exercise in postabsorptive phase B= High-intensity interval exercise in postprandial phase C= Moderate-intensity continuous exercise in postabsorptive phase D= Moderate-intensity continuous exercise in postprandial phase
  Interventions: Other: High-intensity interval exercise performed in postprandial phase; Other: High-intensity interval exercise performed in postabsorptive phase; Other: Moderate-intensity continuous exercise performed in postprandial phase; Other: Moderate-intensity continuous exercise performed in postabsorptive phase
- B/C/D/A (Experimental): A= High-intensity interval exercise in postabsorptive phase B= High-intensity interval exercise in postprandial phase C= Moderate-intensity continuous exercise in postabsorptive phase D= Moderate-intensity continuous exercise in postprandial phase
  Interventions: Other: High-intensity interval exercise performed in postprandial phase; Other: High-intensity interval exercise performed in postabsorptive phase; Other: Moderate-intensity continuous exercise performed in postprandial phase; Other: Moderate-intensity continuous exercise performed in postabsorptive phase
- C/D/A/B (Experimental): A= High-intensity interval exercise in postabsorptive phase B= High-intensity interval exercise in postprandial phase C= Moderate-intensity continuous exercise in postabsorptive phase D= Moderate-intensity continuous exercise in postprandial phase
  Interventions: Other: High-intensity interval exercise performed in postprandial phase; Other: High-intensity interval exercise performed in postabsorptive phase; Other: Moderate-intensity continuous exercise performed in postprandial phase; Other: Moderate-intensity continuous exercise performed in postabsorptive phase
- D/A/B/C (Experimental): A= High-intensity interval exercise in postabsorptive phase B= High-intensity interval exercise in postprandial phase C= Moderate-intensity continuous exercise in postabsorptive phase D= Moderate-intensity continuous exercise in postprandial phase
  Interventions: Other: High-intensity interval exercise performed in postprandial phase; Other: High-intensity interval exercise performed in postabsorptive phase; Other: Moderate-intensity continuous exercise performed in postprandial phase; Other: Moderate-intensity continuous exercise performed in postabsorptive phase

INTERVENTIONS:
Other: High-intensity interval exercise performed in postprandial phase — Exercises were performed on a cycle ergometer (Excalibur Sport, Lode B.V.). Exercise began with a 3-min warm-up at 20% of maximum aerobic power (MAP) and ended with a 2-min active recovery at 20% of MAP. The high-intensity interval exercise protocol consisted of ten 1-min intervals at 100% of MAP, each interspersed with 1-min of passive recovery. For the postprandial state, exercise began 1.5 hours after the start of lunch and the corresponding meal-related bolus/rapid-acting insulin (i.e., in the early afternoon).
Other: High-intensity interval exercise performed in postabsorptive phase — Exercises were performed on a cycle ergometer (Excalibur Sport, Lode B.V.). Exercise began with a 3-min warm-up at 20% of maximum aerobic power (MAP) and ended with a 2-min active recovery at 20% of MAP. The high-intensity interval exercise protocol consisted of ten 1-min intervals at 100% of MAP, each interspersed with 1-min of passive recovery. For the postabsorptive state, exercise began 5 hours after the start of lunch (i.e., in the late afternoon).
Other: Moderate-intensity continuous exercise performed in postprandial phase — Exercises were performed on a cycle ergometer (Excalibur Sport, Lode B.V.). Exercise began with a 3-min warm-up at 20% of maximum aerobic power (MAP) and ended with a 2-min active recovery at 20% of MAP. The moderate-intensity continuous exercise protocol consisted of continuous exercise at 50% of MAP for 20 minutes. For the postprandial state, exercise began 1.5 hours after the start of lunch and the corresponding meal-related bolus/rapid-acting insulin (i.e., in the early afternoon).
Other: Moderate-intensity continuous exercise performed in postabsorptive phase — Exercises were performed on a cycle ergometer (Excalibur Sport, Lode B.V.). Exercise began with a 3-min warm-up at 20% of MAP and ended with a 2-min active recovery at 20% of maximum aerobic power (MAP). The CONT protocol consisted of continuous exercise at 50% of MAP for 20 minutes. For the postabsorptive state, exercise began 5 hours after the start of lunch (i.e., in the late afternoon).

SUMMARY:
This randomized crossover trial examined whether exercise modality (high-intensity interval exercise vs. moderate-intensity continuous exercise) and timing relative to meals (postprandial vs. postabsorptive) influence glycemic responses in physically active adults with type 1 diabetes. Participants completed four cycling sessions matched for total mechanical load, and glucose levels were monitored during exercise and for 24 hours afterward while accounting for dietary intake and insulin administration. The study hypothesized that glycemic responses differ according to both exercise type and prandial state.

DETAILED DESCRIPTION:
Participants were tested at the laboratory during one inclusion visit followed by 4 intervention visits separated by at least 48 hours and 4 weeks maximum. During the inclusion visit, participants completed the YMCA submaximal cycle-ergometer (Excalibur Sport, Lode B.V.) test to estimate maximal aerobic power (MAP), which was then used to determine subsequent exercise workloads. The test started at 25 W (50 rpm), with increasing power outputs derived from the first-stage heart-rate response. The 3-min stages continued until steady-state heart rate achieved 85% of maximal heart rate minus 10 bpm, with a 1-min extension if heart rate varied by >5 beats·min-¹ between minutes 2 and 3. Participants completed questionnaires about physical activity levels, barriers to physical activity, quality-of-life and hypoglycemia awareness. The next four experimental visits in randomized order consisted of the two aerobic exercises (i.e. high-intensity interval exercise, HIIE and moderate-intensity continuous exercise, CONT), each performed under two different prandial conditions, postprandial (PP) and postabsorptive (PA) state. A triaxial accelerometer (ActiGraph, wGT3X-BT, 30 Hz, epoch set at 60 sec) was worn on the hip from wake-up until bedtime for the day before, during and after each experimental visit. Participants were also asked to record the time, type and amount of food consumed, with the option of photographing meals, as well as in case of multiple daily injection doses/timing of insulin (rapid- and long-acting), the 24 hours before, during and after each visit. Exercises were performed on a cycle ergometer (Excalibur Sport, Lode B.V.) and were matched for total mechanical load and total duration. Both exercises began with a 3-min warm-up at 20% of MAP and ended with a 2-min active recovery at 20% of MAP. The HIIE protocol consisted of ten 1-min intervals at 100% of MAP, each interspersed with 1-min of passive recovery. The CONT protocol consisted of continuous exercise at 50% of MAP for 20 minutes. For the postprandial state, exercise began 1.5 hours after the start of lunch and the corresponding meal-related bolus/rapid-acting insulin, (i.e., in the early afternoon). For the postabsorptive state, exercise began 5 hours after the start of lunch, (i.e., in the late afternoon). Participants were instructed to follow their habitual pre-exercise routine and to replicate, as closely as possible, the same lunch and dinner on the days of the experimental visits. The measurements included: oxygen uptake, heart rate, rate of perceived exertion, muscle vasoreactivity during exercise; capillary glycaemia and lactataemia at several time points during exercise; continuous glucose monitoring data from the personal (used in daily life) device of the participants.

ELIGIBILITY:
Inclusion Criteria:

* Between 18 and 60 years of age
* Regular practice of physical activity (at least 2 training sessions/week for at least 3 months)
* Diagnosis of type 1 diabetes for >1 year
* No change in insulin delivery method (i.e., multiple daily injections [MDI], continuous subcutaneous insulin infusion [CSII] in open or closed loop) over the previous 3 months
* Use of a continuous glucose monitoring (CGM) device in daily life

Exclusion Criteria:

* Diabetes-related complications except for background retinopathy

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 21 (Actual)
Dates: Start 2023-02-08 (Actual); Primary Completion 2025-01-17 (Actual); Study Completion 2025-05-09 (Actual)

PRIMARY OUTCOMES:
Capillary glycemia | At rest before exercise, then at 10 and 20 min of exercise, at 2 min of active recovery post-exercise, and at 10 min of passive recovery post-exercise.
  Blood glucose meter

SECONDARY OUTCOMES:
Interstitial glucose | The 24 hours before and the 24 hours after each visit
  Continuous Glucose Monitoring system used by the participant in daily life
Capillary blood lactate | At rest before exercise, then at 10 and 20 min of exercise, at 2 min of active recovery post-exercise, and at 10 min of passive recovery post-exercise.
  Measured using the Lactate Scout device.
Oxygen consumption | During a 5-min rest before exercise, a 3-min warm-up, 20-min of exercise, a 2-min active recovery post-exercise, and a 10-min passive recovery post-exercise.
  Measured with a mask and a Vynthus CPX, Vyaire Medical
Rate of Perveived Exertion | At rest before the exercise, and then at 5-min, 10-min, 15-min and 20-min of exercise, at 2-min active recovery post-exercise and at 5 and 10-min passive recovery post-exercise.
  Rate of Perveived Exertion from the Borg Scale (6 to 20 scale)
Variation of muscle blood volume. | During a 5-min rest before exercise, a 3-min warm-up, 20-min of exercise, a 2-min active recovery post-exercise, and a 5-min passive recovery post-exercise.
  Measured with Near infrared spectroscopy (Artinis, PortaLite)
Heart rate | During a 5-min rest before exercise, a 3-min warm-up, 20-min of exercise, a 2-min active recovery post-exercise, and a 10-min passive recovery post-exercise.
  Measured with Polar V800.
Perceived pleasure | At the end of 10-min passive recovery post-exercise.
  Physical activity enjoyment scale (PACES) 18 items rated on a 7-point Likert scale.

CONTACTS AND LOCATIONS:
Locations (1):
- Unité de Recherche Pluridisciplinaire Sport, Santé, Société (URePSSS - ULR 7369), Loos, France

IPD SHARING:
Plan to Share IPD: Yes
The investigators will share on http://recherche.data.gouv.fr all anonymized data presented in the publication of the results
Time Frame: From the acceptance date of publication
Access Criteria: Access on e-mail request to investigators